CLINICAL TRIAL: NCT03073096
Title: Performing a Lymphatic-venous Anastomosis at Time of Nodal Dissection in Patients Requiring Complete Axillary or Groin Dissection for the Prevention of Lymphedema
Brief Title: LYMPHA: Eliminating the Burden of Lymphedema in Patients Requiring Nodal Dissection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough resources to continue the study especially with Covid-19
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20170146 form 6131
Record Dates: First submitted 2017-02-21; First posted 2017-03-08 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Lymph Node Disease
Keywords: axillary nodal dissection; groin nodal dissection

STUDY DESIGN:
Intervention Model Description: All melanoma and other skin cancers (merkel cell carcinoma, squamous cell carcinoma as well as sarcoma patients requiring a nodal dissection (groin or axillary) will be offered to have a LVA at time of nodal dissection to prevent lymphedema.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Other): LVA at time of nodal dissection
  Interventions: Procedure: LVA at time of nodal dissection

INTERVENTIONS:
Procedure: LVA at time of nodal dissection — Patients will receive a lymphatic-venous anastomosis at time of their required nodal dissection

SUMMARY:
Lymphedema is the build-up of lymph fluid in the body's tissue causing chronic, debilitating swelling. This commonly occurs as a result of a disruption of the lymphatic system during lymph node dissection surgeries. In melanoma patients, the incidence of lymphedema ranges from 5-10% in the arms following an axillary dissection, and 28-40% in the legs following groin dissection. LYMPHA (LYmphatic Microsurgical Preventive Healing Approach) is an innovative microsurgical technique where blocked lymphatic vessels are drained into the blood circulation by surgically creating a shunt between a lymphatic channel and a blood vessel called a lymphatic-venous bypass. Recently, LYMPHA has been shown to prevent lymphedema when performed at the time of nodal dissection. We propose a prospective pilot study evaluating the practice of the LYMPHA technique for the primary prevention lymphedema at The Ottawa Hospital. The novel use of the LYMPHA technique holds the potential to prevent lymphedema rather than to attempt to treat it once it has already progressed and as a result will not only improve the quality of life of the cancer patients, but also decrease health care costs associated with treating lymphedema.

DETAILED DESCRIPTION:
Consenting patients will have the LYMPHA procedure at the time of planned axillary or groin dissection surgery for the prevention of upper and lower extremity lymphedema, respectively. The node dissection will be performed by Dr. Nessim, while the LYMPHA technique will be performed by the plastic surgeon, Dr. Momtazi, trained in microsurgical technique. The LYMPHA procedure consists of performing lymphatic-venous anastomoses (LVA) at the time of the node dissection. Patent blue dye will be injected into the patient approximately 10 minutes before skin incision. This will allow mapping of the lymphatic channels for identification for bypass. The node dissection will then be performed with preservation of the saphenous vein in the leg and the anterior branch of the axillary vein in the axilla. Afferent lymphatic vessels will be sutured into the saphenous vein or a branch of the axillary vein distal to a competent valve, respectively. The total duration of the surgery is approximately 3 hours. The LYMPHA technique accounts for an additional 30 minutes to the standard 2-2.5 hours allocated to the node dissection.

Pre-surgery, patients will have baseline limb circumference measurements of both the surgery-affected and unaffected limbs (arms or legs). Patients will be followed up clinically at every 3 months up to a year, and then again at the end of the second year (at the 24 month-mark only). At each follow-up visit, patients will have a physical examination and their circumferential limb measurements will be taken with measuring tape at three specific intervals up the limb. For example, patients undergoing an axillary dissection will have the circumference of their wrist taken, and then again 4 cm proximal to the wrist, then 8 cm proximal to the wrist, and so forth. The method will be used for the legs but starting at the ankle. Volume will be calculated indirectly, using Dr. Brorson's truncated cone method (13). Patients will also fill out a limb lymphedema-specific quality of life questionnaire (LYMQOL) administered by the Clinical Research Coordinator pre- and post-surgery. Each patient will have a total of 2 years of participation time.

Pre-surgery, patients will have baseline limb circumference measurements of both the surgery-affected and unaffected limbs (arms or legs). Patients will be followed up clinically at every 3 months up to a year, and then again at the second year. At each follow-up visit, patients will have a physical examination and their circumferential limb measurements will be taken with measuring tape at three specific intervals up the limb. Patients will also fill out a limb lymphedema-specific quality of life questionnaire (LYMQOL) administered pre- and post-surgery.

1. Primary Objective: To evaluate the success rate of performing the LYMPHA procedure. Success is defined as a completed LYMPHA procedure i.e. successful LVA.
2. Secondary Objective: To evaluate the feasibility of follow-up assessments i. establish the ability to obtain pre- and post- limb measurements ii. obtain limb-specific quality of life information iii. design a protocol for a randomized controlled trial comparing lymphedema rates in patients receiving a lymphadenectomy + lymphatic-venous bypass versus lymphadenectomy alone.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary melanoma, soft tissue sarcoma, squamous cell carcinoma or merkel cell carcinoma of the trunk or chest.
* Node-positive cancer requiring an axillary or groin lymphadenectomy

Exclusion Criteria:

* Patients receiving a sentinel lymph node biopsy alone
* Patients with a cancer on the upper or lower extremities are excluded (i.e. arms or legs).
* Patients with established preoperative lymphedema
* Patients with post-thrombotic syndrome, peripheral vascular disease
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2020-06-03 (Actual)

PRIMARY OUTCOMES:
Difference in limb volume between surgery-affected and surgery-unaffected limb at baseline, 3, 6, 9, 12 and 24 months | every 3 months up to a year, again at year 2
  At each follow-up visit, patients will have a physical examination and their circumferential limb measurements will be taken with measuring tape at three specific intervals up the limb. For example, patients undergoing an axillary dissection will have the circumference of their wrist taken, and then again 4 cm proximal to the wrist, then 8 cm proximal to the wrist, and so forth. The method will be used for the legs but starting at the ankle. Volume will be calculated indirectly, using Dr. Brorson's truncated cone method.

SECONDARY OUTCOMES:
Limb-lymphedema-specific Quality of life assessment at baseline, 3, 6, 9, 12 and 24 months through the LYMQOL questionnaire | every 3 months up to a year, again at year 2
  Patients will fill out a limb lymphedema-specific quality of life questionnaire (LYMQOL). This includes the LYMQOL-arm or the LYMQOL-leg.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Nessim, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feldman S, Bansil H, Ascherman J, Grant R, Borden B, Henderson P, Ojo A, Taback B, Chen M, Ananthakrishnan P, Vaz A, Balci F, Divgi CR, Leung D, Rohde C. Single Institution Experience with Lymphatic Microsurgical Preventive Healing Approach (LYMPHA) for the Primary Prevention of Lymphedema. Ann Surg Oncol. 2015 Oct;22(10):3296-301. doi: 10.1245/s10434-015-4721-y. Epub 2015 Jul 23. PMID 26202566
- [Background] Boccardo F, Valenzano M, Costantini S, Casabona F, Morotti M, Sala P, De Cian F, Molinari L, Spinaci S, Dessalvi S, Campisi CC, Villa G, Campisi C. LYMPHA Technique to Prevent Secondary Lower Limb Lymphedema. Ann Surg Oncol. 2016 Oct;23(11):3558-3563. doi: 10.1245/s10434-016-5282-4. Epub 2016 May 24. PMID 27221358
- [Background] Morotti M, Menada MV, Boccardo F, Ferrero S, Casabona F, Villa G, Campisi C, Papadia A. Lymphedema microsurgical preventive healing approach for primary prevention of lower limb lymphedema after inguinofemoral lymphadenectomy for vulvar cancer. Int J Gynecol Cancer. 2013 May;23(4):769-74. doi: 10.1097/IGC.0b013e318287a8e8. PMID 23485932
- [Background] Boccardo F, Casabona F, De Cian F, Friedman D, Murelli F, Puglisi M, Campisi CC, Molinari L, Spinaci S, Dessalvi S, Campisi C. Lymphatic microsurgical preventing healing approach (LYMPHA) for primary surgical prevention of breast cancer-related lymphedema: over 4 years follow-up. Microsurgery. 2014 Sep;34(6):421-4. doi: 10.1002/micr.22254. Epub 2014 Mar 26. PMID 24677148
- [Background] Torrisi JS, Joseph WJ, Ghanta S, Cuzzone DA, Albano NJ, Savetsky IL, Gardenier JC, Skoracki R, Chang D, Mehrara BJ. Lymphaticovenous bypass decreases pathologic skin changes in upper extremity breast cancer-related lymphedema. Lymphat Res Biol. 2015 Mar;13(1):46-53. doi: 10.1089/lrb.2014.0022. Epub 2014 Dec 18. PMID 25521197
- [Background] Starritt EC, Joseph D, McKinnon JG, Lo SK, de Wilt JH, Thompson JF. Lymphedema after complete axillary node dissection for melanoma: assessment using a new, objective definition. Ann Surg. 2004 Nov;240(5):866-74. doi: 10.1097/01.sla.0000143271.32568.2b. PMID 15492570
- [Background] Mehrara BJ, Zampell JC, Suami H, Chang DW. Surgical management of lymphedema: past, present, and future. Lymphat Res Biol. 2011;9(3):159-67. doi: 10.1089/lrb.2011.0011. PMID 22066746
- [Background] Gomberawalla A, Feldman S. LYMPHA: New Innovation, Not Old Practice. J Clin Oncol. 2016 Sep 1;34(25):3108-9. doi: 10.1200/JCO.2016.67.8987. Epub 2016 Jun 13. No abstract available. PMID 27298413
- [Background] van Akkooi AC, Bouwhuis MG, van Geel AN, Hoedemaker R, Verhoef C, Grunhagen DJ, Schmitz PI, Eggermont AM, de Wilt JH. Morbidity and prognosis after therapeutic lymph node dissections for malignant melanoma. Eur J Surg Oncol. 2007 Feb;33(1):102-8. doi: 10.1016/j.ejso.2006.10.032. Epub 2006 Dec 11. PMID 17161577
- [Background] Brorson H, Hoijer P. Standardised measurements used to order compression garments can be used to calculate arm volumes to evaluate lymphoedema treatment. J Plast Surg Hand Surg. 2012 Dec;46(6):410-5. doi: 10.3109/2000656X.2012.714785. PMID 23157502
- [Background] Boccardo FM, Casabona F, Friedman D, Puglisi M, De Cian F, Ansaldi F, Campisi C. Surgical prevention of arm lymphedema after breast cancer treatment. Ann Surg Oncol. 2011 Sep;18(9):2500-5. doi: 10.1245/s10434-011-1624-4. Epub 2011 Mar 3. PMID 21369739